CLINICAL TRIAL: NCT00341341
Title: Impact of a Patient's Lung Cancer Diagnosis on Relatives' Understanding of Genetic Risk Information and Receptivity to Quit Smoking
Brief Title: Impact of Lung Cancer Diagnosis on Relatives' Understanding of Genetic Risk and Receptivity to Quit Smoking
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905054; 05-HG-N054
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-16

CONDITIONS: Lung Cancer
Keywords: Smoking; Smoking Cessation; GSTM1; Glutathione S. Transferase; Lung Cancer; Smokers; Genetic Risk Communication
MeSH Terms: conditions — Lung Neoplasms; Smoking; Smoking Cessation

SUMMARY:
This study will explore beliefs and knowledge about genetics and smoking among smokers who have a first or second degree relative with advanced lung cancer, and whether their understanding of genetic risk influences their desire to quit smoking.

Healthy adult smokers between 18 and 55 years of age who are first or second degree relatives (e.g., siblings, children, grandchildren, nieces, nephews, grandnieces or grandnephews) of a patient with advanced lung cancer who is receiving care at the Moffitt Cancer Center and Research Institute in Tampa, Fla. and the GUMC/LCCC, may be eligible for this study. Participants must be able to complete computer online surveys.

Participants log on to a password-protected website to complete online educational sessions and surveys. The educational sessions include information on: 1) the role of smoking and genetics in the development of lung cancer; 2) glutathione S transferase (GSTM1), an enzyme made by the GSTM1 gene that "cleans up" toxins such as cigarette smoke and that may play a role in preventing lung cancer from developing; 3) pros and cons of being tested for GSTM1; and 5) a series of questions and answers about genetic testing. Participants are offered free genetic testing for GSTM1, and those who wish to be tested are sent materials to collect a sample from inside the cheek using a mouth rinse and return it to a laboratory at Duke University Medical Center. They later receive their results online.

Participants also complete online surveys that ask about their risk perceptions, beliefs and attitudes related to lung cancer, emotional responses to their relative's diagnosis, smoking history and motivation to quit, reactions to information about smoking and genetic risk, and interest in receiving smoking cessation services. They are asked to review depictions and descriptions of smoking cessation materials offered through a quit smoking program at Duke University Medical Center and to evaluate the extent to which the various materials might be helpful. They are offered additional information among categories they can choose from.

Participants are surveyed again by telephone 6 months after completing the online surveys.

DETAILED DESCRIPTION:
The overarching objective of this observational prospective "Genetic Risk & Lung Cancer Study" is to evaluate the impact of a loved one's lung cancer diagnosis on relative's seeking and processing of information related to risks of smoking, genetic susceptibility, and their receptivity to smoking cessation services. We plan to recruit 150 relatives of lung cancer patients who are receiving care at H. Lee Moffitt Cancer Center and Research Institute in Tampa, Florida and the Lombardi Comprehensive Cancer Center at the Georgetown University Medical Center (GUMC/LCCC). First- or second-degree blood relatives who are current smokers between the ages of 18 to 55 will be eligible for the study. Because these relatives will be living throughout the United Sates, a web-based research protocol will be employed. A nurse recruiter will approach patients at Moffitt and assess their willingness to do a telephone survey The overarching objective of this observational prospective "Genetic Risk & Lung Cancer Study" is to evaluate the impact of a loved one's lung cancer diagnosis on relative's seeking and processing of information related to risk of smoking, genetic susceptibility, and their receptivity to smoking cessation services. We plan to recruit 150 relatives of lung cancer patients who are receiving care at H. Lee Moffitt Cancer Center and Research Institute in Tampa, Florida. First-or second-degree relatives who are current smokers between the ages 18 to 55 will be eligible for the study. Because these relatives will be living throughout the United States, a web-based research protocol wil be employed. A nurse recruiter will approach patients at Moffitt and assess their willingness to do a telephone survey to enumerate their relatives who smoke and be asked to give permission to contact none, some or all of these relatives. These survey contacts with patients and contacts with relatives for screening and recruitment will be conducted in partnership with an ongoing recruitment activities for a five-year, NCI-funded randomized controlled intervention trial (RCT) at Duke University Medical Center (Quit Smoking Program for Lung Cancer Patient's Families or "Family Ties", Duke IRB# 4620, Bastian, PI). Relatives who agree to participate will be asked to log on to a password protected website and view two online educational sessions and complete three online surveys. As part of the educational session, participants will be offered free geneticsusceptibility testing for glutathione S transferase (GSTM1). Participants who accept testing will receive their result online. Participants who decline testing will be retained in the the study and offered all the same smoking cessation services provided to those who accept testing. Participants will be sent instructions to collect their own buccal samples and postage-paid mailing envelopes to return the sample to a CLIA-approved laboratory at Duke. Survey assessments will include questions about risk perceptions, beliefs and attitudes related to lung cancer, emotional responses to the patient's diagnosis, smoking history, motivation to quit, reactions to information about smoking and genetic risk, interest in genetic testing, comprehension of susceptibility feedback, and interest in receiving smoking cessation services. The primary outcome variable will be seeking of free quit smoking services. Participating relatives will be surveyed by telephone via the Duke RCT infrastructure 6-months after completing the online protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

The target sample for the study is healthy adult smokers ages 18 to 55 who are first or second degree blood relatives (e.g., siblings, sons, daughters, grandsons, granddaughters, nieces, nephews, grandnieces, grandnephews) of a late stage lung cancer patient (Stage IIIB or IV) who is receiving care at MCC.

Aside from age and blood relationship to the lung cancer patient, eligibility criteria also will include the following:

No current or previous diagnosis of cancer;

Has access and some willingness to use the internet;

Is willing to be contacted by NIH study staff;

Has a score lower than 14 on the Centers for Epidemiological Survey of Depression (CESD);

Is English speaking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 757 (Estimated)
Dates: Start 2004-12-07; Study Completion 2010-07-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alexandrie AK, Nyberg F, Warholm M, Rannug A. Influence of CYP1A1, GSTM1, GSTT1, and NQO1 genotypes and cumulative smoking dose on lung cancer risk in a Swedish population. Cancer Epidemiol Biomarkers Prev. 2004 Jun;13(6):908-14. PMID 15184245
- [Background] Aspinwall LG, Taylor SE. Effects of social comparison direction, threat, and self-esteem on affect, self-evaluation, and expected success. J Pers Soc Psychol. 1993 May;64(5):708-22. doi: 10.1037//0022-3514.64.5.708. PMID 8505703
- [Background] Belogubova EV, Togo AV, Karpova MB, Kuligina ESh, Buslova KG, Ulibina JM, Lemehov VG, Romanenko SM, Shutkin VA, Hanson KP, Hirvonen A, Imyanitov EN. A novel approach for assessment of cancer predisposing roles of GSTM1 and GSTT1 genes: use of putatively cancer resistant elderly tumor-free smokers as the referents. Lung Cancer. 2004 Mar;43(3):259-66. doi: 10.1016/j.lungcan.2003.08.019. PMID 15165083